CLINICAL TRIAL: NCT05625555
Title: Clinical Predictors of Intravenous Ketamine Response in Treatment-Resistant Depression: A Randomized, Double-Blind, Midazolam-Controlled Pilot Study
Brief Title: Predictors of Intravenous Ketamine Response in TRD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abraham Nunes (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Abraham Nunes, Psychiatrist/Assistant Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DALKETCLIN
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder; Bipolar Disorder
Keywords: Treatment Resistant Depression; Major Depressive Disorder; Bipolar Disorder; Clinical Prediction; Ketamine; Midazolam
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Participants will receive either a single infusion of IV Ketamine (KET; 0.5mg/kg over 40 minutes) or Midazolam (MID; 30μg/kg over 40 minutes). Investigators will randomize infusion sequences in a 1-to-1 ratio: KET followed by MID or vice versa. Infusions will be administered on Day 0 and Day 21, separated by a 20-day washout period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants will be randomly assigned to receive Ketamine or Midazolam
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Participants will receive either Ketamine or Midazolam based on what they initially received
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — IV Ketamine infusion 0.5mg/kg over 40 minutes
  Other Names: Ketamine Hydrochloride; Kevlar
  Arms: Ketamine
Drug: Midazolam — IV Midazolam infusion 30μg/kg over 40 minutes
  Other Names: Midazolam Hydrochloride
  Arms: Midazolam

SUMMARY:
For patients with treatment-resistant depression (TRD), a single low dose of intravenous (IV) ketamine can help relieve symptoms as quickly as 24 hours later.

The main problem with IV ketamine for TRD is that the effect is short-lived, lasting only days to 1 or 2 weeks. Furthermore, IV ketamine is a resource-intensive treatment, and the safety of long-term, repeated use for depression is unknown. To provide this treatment in a safe and cost-effective way, Investigators must allocate it efficiently to those patients who have the greatest need and probability of benefit. Therefore, this project aims to find clinical features (signs, symptoms, and parts of a patient's history) that will help predict which patients are most likely to respond to a single dose of IV ketamine for TRD. This will help guide patient selection and triaging.

Investigators will recruit 40 participants with TRD over one year, and randomize them to one of two conditions (ketamine followed by an active placebo 3-weeks later, or vice versa). With clinical data collected through detailed interviews, questionnaires, actigraphy, speech sampling, electroencephalography (EEG), and computerized tasks, this study design will let us evaluate how well such factors predict (A) rapid response at 24-hours, and (B) sustained response at 7 and 14 days.

DETAILED DESCRIPTION:
Study Design:

This will be a randomized, double-blinded, midazolam-controlled crossover trial. There is no perfect control agent for studies of subanaesthetic IV ketamine, but midazolam is generally thought to be superior to normal saline since it is not an antidepressant, yet is psychoactive and thus should better preserve blinding. Participants will undergo psychiatric assessment to establish diagnosis and determine suitability. After providing informed consent for participation, participants will wear a GENEActive accelerometer on the non-dominant wrist for the duration of the trial, beginning 21 days prior to the first infusion. Participants will complete a set of rating scales, anhedonia measures and computerized tasks. On Day 0 (infusion day), participants will receive either a single infusion of IV ketamine (KET) (KET; 0.5mg/kg over 40 minutes) or midazolam (MID) (MID; 30μg/kg over 40 minutes) diluted in 0.9% NaCl by an intravenous pump. Investigators will randomize infusion sequences in a 1-to-1 ratio: KET followed by MID (K→M) or vice versa (M→K). Infusions will be administered on Days 0 and 21, separated by a 20-day washout period. This duration balances the need to establish comparable baselines at each crossover phase and the ethical consideration of not allowing depressive symptoms to remain untreated for an unreasonable amount of time.

Investigators will obtain objective depression ratings with the Montgomery-Åsberg Depression Rating Scale (MADRS) on Days -1, 1, 7, 14, 20, 22, 28, 35, and 41. Participants will provide weekly self-ratings of depressive symptoms (using the Quick Inventory of Depressive Symptoms 16-item self-rated version; QIDS 16-SR). Weekly symptom monitoring will continue for 20 days following the second infusion. Anhedonia will be measured using both self-reported rating scale measures as well as behavioural task. Patients will provide self-ratings using the Snaith-Hamilton Pleasure Scale - 14 items (SHAPS), the Dimensional Anhedonia Rating Scale - 17 items (DARS), and Positive Valence System Scale - 21 items (PVSS-21). Several aspects of subjective sleep and circadian rhythms will be measured via self-report questionnaires. The Pittsburgh Sleep Quality Index (PSQI) will measure general sleep quality and sleep disturbance, and the Basic Language Morningness Scale (BALM) will be used to measure subjective chronotype (morningness-eveningness) of patients. Both will be completed by participants prior to the first infusion and 14 days after each infusion.

Participants will complete the Epworth Sleepiness Scale (ESS) to measure daytime sleepiness symptoms, as well as the Fatigue Scale Severity Scale (FSS) to measure symptoms of fatigue. Both ESS and FSS will be completed the day before and after each infusion, and every 7 days.

Study Groups:

Participants will receive either (A) 0.5mg/kg of ketamine hydrochloride or (B) 30μg/kg of MID diluted in 0.9 percent Sodium chloride (NaCl) over 40 minutes by an intravenous pump. The KET and MID doses are similar to those used in previous studies, and selected to minimize the possibility of unblinding. Participants must abstain from consuming grapefruit juice or benzodiazepines for 24 hours preceding the infusion since the former is a potent CYP3A4 inhibitor that may reduce the rate of midazolam and ketamine elimination, and the latter reduces the response to ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Able to fluently read in English with or without optical correction
* Ability to understand and comply with the study requirements

  * This is determined by the investigators
* Provision of written informed consent
* Documented diagnosis of MDD or bipolar disorder meeting DSM-5 criteria (as confirmed by the Diagnostic Assessment Research Tool), currently in a single or recurrent episode without psychotic features
* Failure of at least two antidepressant medications from different pharmacological classes, as well as at least one augmentation agent, each of which must have been given at adequate doses for at least 6 weeks (recorded using the Antidepressant Treatment History Form - Short Form).

  * Augmentation strategies include those listed in the 2016 Canadian Network for Mood and Anxiety Treatments (CANMAT) depression guidelines, including a 12-week course of cognitive behavioural therapy or interpersonal therapy.
* MADRS score of ≥25 at initial assessment and Day -1, and no more than 20% improvement between those visits.
* For premenopausal females who are currently sexually active with male partners:

  * Negative urine pregnancy test at enrolment
  * AND commitment to using an appropriate birth control method of their choice throughout the duration of the study, including

    * Intrauterine device
    * Oral contraceptive
    * Long-term injectable contraceptive
    * Double-barrier method
    * Implant
    * Dermal contraception
    * Tubal ligation
* Abstinence from grapefruit juice consumption on the day of infusion
* Abstinence from benzodiazepine use within 24 hours of infusion
* Adherence to maintaining current antidepressant management

Exclusion Criteria:

* Pregnant or breastfeeding
* Allergies to ketamine or midazolam
* Concomitant use of medications with the potential for clinically significant interactions with either ketamine or midazolam (e.g., monoamine oxidase inhibitors, methylene blue)
* Substance related exclusion criteria:

  * Concomitant use of naltrexone or narcotics
  * Positive urine drug screen or history of DSM-5 substance use disorder (except caffeine or nicotine)
  * Previous or current benzodiazepine abuse history
* Psychiatric exclusion criteria:

  * Previous ketamine use (therapeutic or recreational)
  * History of electroconvulsive therapy
  * Comorbid DSM-5 personality disorder with a major impact on mental status
  * Secondary depressive disorders

    * E.g. secondary to stroke, cancer, or other somatic pathology
  * Subjects who will be starting psychotherapy during the trial period, or have only recently started psychotherapy within 2 months of the trial
* Medical comorbidity related exclusion criteria:

  * Evidence on history or chart review of any of the following:

    * Epilepsy
    * Any current or historical occurrence of renal disease

      * Clinically significant abnormalities of liver function tests (total bilirubin, albumin, prothrombin time and international normalized ratio [PT/INR], gamma-glutamyl transferase [GGT], alkaline phosphatase [ALP]). Clinical significance of any abnormal liver function tests will be evaluated by the study anesthesiologists. Patients with clinically significant abnormalities suggesting hepatic disease will be excluded.
      * Liver enzymes (AST, ALT) three times the upper normal limit at screening
      * Exception: of history of acute kidney injury or transient reductions in glomerular filtration rate that have fully resolved for at least three months
    * Any current or historical occurrence of hepatic disease

      * Abnormal liver function tests
      * Liver enzymes three times the upper normal limit at screening
      * Exception: History of transient elevations of liver enzymes or reduction in liver function that have re-normalized for the past three months (as per criteria above concerning function/enzymes)
    * Myocardial infarct within a year prior to initial randomization
    * Chronic obstructive pulmonary disease
    * Untreated obstructive sleep apnea
    * Cerebrovascular disease (including history of cerebrovascular accident)
    * Intracerebral structural lesions
    * Viral hepatitis B or C
    * Acquired immunodeficiency syndrome
    * Interstitial cystitis
    * Glaucoma
    * Uncontrolled hypertension
    * Decompensated heart failure
  * Current uncorrected thyroid pathology or recent correction within 30 days (correction of thyroid function for longer than 1 month is admissible).
  * Any unstable somatic pathology or clinically significant investigational abnormality (biochemical, ECG) that investigators believe would be negatively impacted by study procedures or that would negatively impact study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery Åsberg Depression Rating Scale Score | 24 hours, 7 days, 14 days, 20 days
  Montgomery Åsberg Depression Rating Scale (MADRS) measures depressive symptoms. The scores for each item ranges from 0 to 6 and total scores range from 0 to 60, with higher scores indicating more severe depression. Researchers will investigate the degree to which each clinical feature predicts Days 1, 7, 14, and 20 post-infusion MADRS using a biomarker prediction model.

SECONDARY OUTCOMES:
Weekly self-ratings of Generalized Anxiety Disorder 7 Scale | 24 hours, 7 days, 14 days, 20 days
  Generalized Anxiety Disorder 7 Scale (GAD-7) measures symptoms of anxiety. The scores for each item ranges from 0 to 3, and total scores range from 0 to 21 with higher scores indicating more severe anxiety. Researchers will investigate the degree to which clinical features predict change in participants' GAD-7 score.
The Snaith-Hamilton Pleasure Scale | 24 hours, 20 days
  Researchers will investigate change in anhedonic symptoms after treatment based on total scores from the Snaith-Hamilton Pleasure Scale (SHAPS), which is a 14-item scale that measures anhedonia. Final scores range from 0-14 with higher scores indicates higher levels of anhedonia.
Dimensional Anhedonia Rating Scale | 24 hours, 20 days
  Researchers will investigate change in anhedonic symptoms after treatment using the Dimensional Anhedonia Rating Scale (DARS). It is a 17-item scale that measures desire, motivation, effort and consummatory pleasure across four reward-related domains. Scores ranges from 0 to 68 with higher values indicating less anhedonia.
The Positive Valence Systems Scale | 24 hours, 20 days
  Researchers will investigate change in anhedonic symptoms after treatment based on the total scores from the Positive Valence Systems Scale (PVSS-21). It is a 21-item scale that measures fine-grained details of hedonic capacity.
Probabilistic Reward Task | 24 hours after each infusion, 20 days after each infusion
  Researchers will evalute change in anhedonic symptoms after treatment using the Probabilistic Reward Task is a neurocognitive computerized task that objectively measures the degree to which the patient can modulate behavior based on reward. 3 Blocks of 100 trials each are separated by thirty-second breaks. A short (11.5 mm) or Long (13 mm) mouth then appears for 100 ms, after which subjects are given a maximum of 7900 ms to indicate whether the mouth presented was short or long by pressing either the left or right shift key.
  In each block, short and long mouth stimuli are shown 50 times each. The central feature of this task is that correct responses are asymmetrically rewarded. That is, for any given task administration, either the long or short mouth is designated as "rich," and the other "lean." Correct classification yields a reward 75% of the time for the "rich" stimulus, but only 30% of the time for the "lean" stimulus.
Fatigue Severity Scale | 24 hours, 7 days, 14 days, 20 days
  Researchers will evaluate the effects of ketamine on change in sleep and circadian function based on Fatigue Severity Scale (FSS) is a 9-item scale that measures symptoms of fatigue. The items are scored on a 7 point scale with 1 for strongly disagree and 7 for strongly agree. The higher the score, the greater the fatigue severity.
Epworth Sleepiness Scale | 24 hours, 7 days, 14 days, 20 days
  Researchers will investigate the effects of ketamine on change in sleep and circadian function based on the Epworth Sleepiness Scale (ESS). It is an 8-item scale that measures daytime sleepiness symptoms. Total scores range from 0 to 24 with higher scores representing higher levels of excessive daytime sleepiness.
Basic Language Morningness Scale | 24 hours, 7 days, 14 days, 20 days
  Researchers will investigate the effects of ketamine on change in sleep and circadian function based on theBasic Language Morningness Scale (BALM), which is a 13-item scale that measures subjective chronotype (morningness-eveningness). Total scores range from 16 to 86, scores of 41 and below indicate "evening types" scores of 42-58 indicate "intermediate types" and scores of 59 and above indicate "morning types".

OTHER OUTCOMES:
Migraine Severity Questionnaire | 7 days
  The scores for some items range from 0 to 4 and others from 0 to 3, and total scores range from 4 to 15, with higher scores indicating more severe migraine. As an exploratory outcome, researchers will investigate the degree to which ketamine infusions affect migraine symptoms, and whether changes in migraine severity are associated with depressive symptom improvements.
Measures of psychomotor behaviour to predict depressive severity | 14 days before the first infusion, 7 days before the first infusion, 1 day before the first infusion, day of the infusions, 24 hours, 7 days, 20 days after each infusion
  Participants will wear an actigraphic device throughout the study and they will provide speech samples on Days -1, 1, 20, 22 and 41.
  Researchers will determine whether measures of psychomotor behaviour (actigraphy and speech) can be used to predict depressive severity. For these analyses, the outcome measures will be MADRS scores at Days -14, -7, -1, 1, 7, 14, 20, 22, 28, 35, and 41.
Effect of treatment on mnemonic discrimination performance in depression | 24 hours before the infusions, 24 hours after the infusions, 20 days after the infusions.
  The Mnemonic Similarity Task (MST) is a behaviour observed during recognition memory tasks, in which individuals are required to distinguish novel stimuli from those that have previously been observed during an econding plase (OLD stimuli). When a novel stimulus is highly similar to an OLD one, people with poor mnemonic discrimination have a higher probability of falsely classifying the novel stimulus as old. That is, poor mnemonic discrimination is essentially the susceptibility of one's memory to interference arising from the similarity between stimuli/events, regardless of overall recognition memory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Nunes, MD PhD MBA FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Mood Disorders Program, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided